CLINICAL TRIAL: NCT07305727
Title: Developing a Radiomic MRI Model Predictive of Response to Concomitant Chemoradiotherapy in Locally Advanced Cervical Cancer. A Prognostic, Retrospective, Open-label, Multicenter, Descriptive and Analytical Clinical Cohort Study
Brief Title: A Radiomic MRI Predictive Model for Response to Concomitant Chemoradiotherapy in Locally Advanced Cervical Cancer
Acronym: EPICOL-R
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: SIRIC/2024/FF01
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Uterine Cervical Neoplasms; Cervical Cancer by FIGO Stage 2018
Keywords: cancer; cervix; survival modeling; radiomic models
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cervical cancer is the fourth most common cancer in women worldwide, with approximately 604,000 new cases in 2020.Treatment for locally advanced cervical cancer is based on a combination of radiotherapy and chemotherapy. The response to concomitant chemoradiotherapy vary from one woman to another. Predicting the response to these treatments would allow early consideration of alternative therapies for patients identified as less responsive to standard treatments. A 5-year recurrence-free survival is approximately 79% for stages IB and IIA and 59% for stages III and IVA, with approximately 36% of local failures despite chemoradiotherapy. In a few studies,the radiomic MRI approach in locally advanced cervical cancers has shown to be prognostic for locoregional recurrence or survival but these models still need to be explored and validated.The EPICOL cohort, a clinical-biological cohort of 136 patients treated with chemoradiotherapy for locally advanced cervical cancer at the Montpellier Cancer Institute or Nîmes University Hospital, will be used to develop a predictive model of response to chemoradiotherapy based on radiomic data from pelvic MRIs before and after treatment.

DETAILED DESCRIPTION:
Cervical cancer is an invasive cancer that develops from the squamous epithelium of the cervix. Worldwide, cervical cancer is the fourth most common cancer in women, with approximately 604,000 new cases in 2020.Treatment for locally advanced cervical cancer (FIGO stage IB3 to IVA) is based on a combination of radiotherapy and chemotherapy (cisplatin 40 mg/m2 x5 or 6 or carboplatin area under the curve 2 if cisplatin is contraindicated). Responses to concomitant chemoradiotherapy remain highly heterogeneous from one woman to another, and predicting the response to these treatments would allow early consideration of alternative therapies for patients identified as less responsive to standard treatments. Indeed, 5-year recurrence-free survival is approximately 79% for stages IB and IIA and 59% for stages III and IVA, with approximately 36% of local failures despite chemoradiotherapy.

The radiomic MRI approach in locally advanced cervical cancers has shown in a few studies to be prognostic for locoregional recurrence or survival. However, these models still need to be explored and validated before they can be implemented in routine clinical practice.

The EPICOL cohort is a clinical-biological cohort of 136 patients treated with chemoradiotherapy for locally advanced cervical cancer at the Montpellier Cancer Institute or Nîmes University Hospital.

The aim is to develop a predictive model of response to chemoradiotherapy based on radiomic data from pelvic MRIs before and after treatment from the EPICOL cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with exclusive radio-chemotherapy for locally advanced cervical cancer (stage Ib-IVb according to the FIGO classification).
* Patients with a minimum of 2 years of post-treatment follow-up.
* Patients for whom the initial biopsy specimen (prior to treatment) is available.
* Patients who have not expressed their opposition to participating in the study.
* Patients who are affiliated with or beneficiaries of a health insurance plan.

Exclusion Criteria:

* Patients under judicial protection, guardianship, or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Human beings who possess a uterus with a cervix.
Study Population: For this study, data from 120 patients for whom we have MRI data from the EPICOL cohort (136 patients included) will be used.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of a magnetic resonance imaging radiomic model on progression-free survival in patients treated for locally advanced cervical cancer. | Month 24
  Time from diagnosis to death from any cause or progression (according to RECIST v1.1 criteria) at 24 months of follow-up.

SECONDARY OUTCOMES:
Prognostic role of an magnetic resonance imaging radiomic model on overall survival in patients treated for locally advanced cervical cancer. | Month 24
  Time between treatment initiation and death from any cause at 24 months of follow-up.
Correlation between the radiomic magnetic imaging radiomic model and Programmed cell Death protein 1 (PD-L1) expression. | Month 24
  Collection of Programmed cell Death protein 1 (PD-L1) expression levels from biopsies from the EPICOL cohort.
Correlation between the radiomic magnetic resonance imaging model and tumor-infiltrating lymphocytes (TILs). | Month 24
  Collection of tumor-infiltrating lymphocyte (TIL) expression levels in biopsies from the EPICOL cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Nimes University Hospital, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pang SS, Murphy M, Markham MJ. Current Management of Locally Advanced and Metastatic Cervical Cancer in the United States. JCO Oncol Pract. 2022 Jun;18(6):417-422. doi: 10.1200/OP.21.00795. Epub 2022 Mar 14. PMID 35286157
- [Background] Zola P, Fuso L, Mazzola S, Piovano E, Perotto S, Gadducci A, Galletto L, Landoni F, Maggino T, Raspagliesi F, Sartori E, Scambia G. Could follow-up different modalities play a role in asymptomatic cervical cancer relapses diagnosis? An Italian multicenter retrospective analysis. Gynecol Oncol. 2007 Oct;107(1 Suppl 1):S150-4. doi: 10.1016/j.ygyno.2007.07.028. Epub 2007 Sep 14. PMID 17868785
- [Background] Autorino R, Gui B, Panza G, Boldrini L, Cusumano D, Russo L, Nardangeli A, Persiani S, Campitelli M, Ferrandina G, Macchia G, Valentini V, Gambacorta MA, Manfredi R. Radiomics-based prediction of two-year clinical outcome in locally advanced cervical cancer patients undergoing neoadjuvant chemoradiotherapy. Radiol Med. 2022 May;127(5):498-506. doi: 10.1007/s11547-022-01482-9. Epub 2022 Mar 24. PMID 35325372
- [Background] Bizzarri N, Russo L, Dolciami M, Zormpas-Petridis K, Boldrini L, Querleu D, Ferrandina G, Pedone Anchora L, Gui B, Sala E, Scambia G. Radiomics systematic review in cervical cancer: gynecological oncologists' perspective. Int J Gynecol Cancer. 2023 Oct 2;33(10):1522-1541. doi: 10.1136/ijgc-2023-004589. PMID 37714669
- [Background] Halle MK, Hodneland E, Wagner-Larsen KS, Lura NG, Fasmer KE, Berg HF, Stokowy T, Srivastava A, Forsse D, Hoivik EA, Woie K, Bertelsen BI, Krakstad C, Haldorsen IS. Radiomic profiles improve prognostication and reveal targets for therapy in cervical cancer. Sci Rep. 2024 May 17;14(1):11339. doi: 10.1038/s41598-024-61271-4. PMID 38760387
- [Background] Li H, Zhu M, Jian L, Bi F, Zhang X, Fang C, Wang Y, Wang J, Wu N, Yu X. Radiomic Score as a Potential Imaging Biomarker for Predicting Survival in Patients With Cervical Cancer. Front Oncol. 2021 Aug 16;11:706043. doi: 10.3389/fonc.2021.706043. eCollection 2021. PMID 34485139